CLINICAL TRIAL: NCT04723693
Title: An Exploration of the Impact of Emicizumab on the Lives of People With Haemophilia and Inhibitors and Their Families
Acronym: EmiandMe
Status: Completed | Type: Observational
Sponsor: Haemnet (Other)
Collaborators: Roche Chugai (Industry)
Responsible Party: Sponsor
Other Study IDs: v4 4Nov2019
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia A With Inhibitor
Keywords: Haemophilia, Quality of Life
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- individuals With Haemophilia A and with inhibitors on emicizumab: Qualitative interviews
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — A single one hour semi structured qualitative interview

SUMMARY:
This study aims to examine the real-life experience and impact of using emicizumab in a cohort of patients with haemophilia and inhibitors, who were prescribed emicizumab as part of the early access to medicine schema (EAMS),those who have been in clinical trials and those now receiving emicizumab as part of routine haemophilia care.

The Investigators also intend to capture the impact of emicizumab use on the lives of close family members (parents/carers/children/partners/siblings). Each participant and his family members will be deemed a study 'dyad'.

This is a prospective, observational cohort qualitative research study to be conducted among patients using emicizumab in routine clinical practice.

The study is designed to allow English-speaking patients and their families to tell their own life stories through narrative accounts. The narratives represent a true sharing of experiences and therefore offers insight into how these patients and families cope with haemophilia.

DETAILED DESCRIPTION:
Emicizumab offers patients protection from bleeding with fewer injections, this should reduce treatment burden. While patient expectation is high (as evidenced by the conversations on UK haemophilia social media sites) there are risks that patients may forget to treat and thus experience bleeds. During clinical trials participants have been monitored closely and, through questionnaire completion, have described improvement in quality of life [Mancuso et al, 2018, Oldenburg et al 2019].

What is also apparent to clinical teams is the dramatic change to life experience of not just the patient but his family - the ability to travel, to plan attending events knowing that bleeds will not occur, even potentially to have another child because of the reduction in treatment burden, particularly the time needed for treatment and rehabilitation.

This therapy represents a substantial shift in the entire life experience of living with and managing haemophilia with inhibitors. As such, there is a need to look beyond the quantitative data collected in clinical trials and to assess the real impact of therapy on the everyday lives of patients and their families, gathered using qualitative research techniques.

Emicizumab has been available in the UK in clinical trials and as part of an Early Access to Medicines Scheme (EAMS) for non-trial eligible patients since spring 2018. It was recently licensed in the UK and is now available for routine clinical care for any person with haemophilia A and an inhibitor.

We hypothesise that patients and their carers/families will be excited about this new treatment option and that for most, if not all, the promise of improved care and quality of life will be a reality.

ELIGIBILITY:
Inclusion Criteria:

* Males
* A diagnosis of Haemophilia A with inhibitors
* Using emicizumab (prescribed by treating clinicians) in usual clinical care.

Exclusion Criteria:

* No history of a Factor VIII inhibitor
* Not currently being treated with emicizumab,
* Does not speak English (for the interviews)
* Does not consent to take part.

Ages: 8 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male participants with Hameophilia A and inhibitors currently on emicizumab prophylaxis and a member of their family
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon P Fletcher, MA, Principal Investigator — Researcher
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher S, Jenner K, Holland M, Khair K. The lived experience of a novel disruptive therapy in a group of men and boys with haemophilia A with inhibitors: Emi & Me. Health Expect. 2022 Feb;25(1):443-454. doi: 10.1111/hex.13404. Epub 2021 Dec 8. PMID 34878209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants will be people with inhibitors using emicizumab (prescribed by treating clinicians) in usual clinical care. Family members of participants will also be included.
Pre-assignment Details: Individual participants and a family member (if available and consented) were interviewed as a dyad pair.
  Individual participants with no available family member were interviewed on their own
Groups:
- Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members: Qualitative interviews
  Qualitative Interview: A single one hour semi structured qualitative interview
Period: Overall Study
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members
Started | 30 (30 participants were recruited in total. * 16 people with haemophilia and inhibitors * 14 family members)
Completed | 28 (28 participants completed the study * 16 people with haemophilia and inhibitors * 12 family members 2 family members withdrew prior to interview Therefore 12 dyad interviews and 4 individual interviews were carried out)
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 16 people with haemophilia and inhibitors and 12 family members
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Reduction in the Burden of the Condition Including Treatment Burden, Bleed Frequency, Pain, Control, Freedom and Missed Opportunities)
Description: To capture the individual participant's and his family's experience of using emicizumab for haemophilia inhibitor therapy and see if there is any reduction in the burden of the condition.
Time Frame: Each participant & family member will take part in a 1 hour semi structured qualitative interview where experiences of his condition, previous treatment & current treatment with emicizumab will be discussed & thematically analysed and reported.
Population: 16 People with Haemophilia and inhibitors were interviewed 12 with family members 14 interviews took place online, one by telephone and one in person. 6 themes emerged: bleeds; pain; treatment burden; control; freedom (for both PwHi and family members) and missed potential.
Measure: Number; unit: participants
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members
Number analyzed (Participants) | 28
participants
  Bleeds | 19
  Pain | 10
  Treatment Burden | 12
  Control | 9
  Freedom | 9
  Missed Opperyunities | 2

2. Secondary Outcome: Treatment Satisfaction (Do the Participants and Their Family Feel That the Change in Treatment Improved Their Condition Control and in What Ways)
Description: To describe patient satisfaction with injections including frequency and numbers of injections, how to remember treatment dates, treatment comfort, bleed rate post switching.
Time Frame: as for outcome 1
Population: People with haemophilia and inhibitors and their family members
Measure: Number; unit: participants
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab
Number analyzed (Participants) | 28
participants
  Treatment Burden | 9
  Control | 9
  Freedom | 9

3. Secondary Outcome: Treatment Expectations
Description: To understand user's expectations of emicizumab and how they see future haemophilia care (less frequent injections, impact on home storage, number of bleeds, reduced hospitalisations etc).
Time Frame: as for outcome 1
Population: people with haemophilia and inhibitors and their family members
Measure: Number; unit: participants
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members
Number analyzed (Participants) | 28
participants
  Increased sense of opportunity on new treatment | 26
  No improvement in opportunities | 2
Statistical Analysis 1: Comparison: Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members; Test type: Other; This is a qualitative interview study and as such no statistical analysis was carried out

4. Secondary Outcome: Treatment Impact
Description: To describe the impact of the change in treatment on the extended family
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members
Number analyzed (Participants) | 12
participants
  Increased control | 6
  Increased freedom | 6
Statistical Analysis 1: Comparison: Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members; Test type: Other; This is a qualitative interview study and as such no statistical analysis was carried out

ADVERSE EVENTS:
Time Frame: Over the course of the 1 hour interview
Arm/Group | Individuals With Haemophilia A and With Inhibitors on Emicizumab and Family Members
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT04723693/Prot_000.pdf